CLINICAL TRIAL: NCT05864807
Title: Safety and Performance of UCon for the Treatment of the Symptoms of Faecal Incontinence (FI) - An Early Feasibility Study
Brief Title: UCon Treatment of the Symptoms of Faecal Incontinence (FI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InnoCon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES_FEAS_01
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Faecal Incontinence; Faecal Incontinence With Faecal Urgency
Keywords: Faecal Incontinence; Faecal Urgency; Neurostimulation; Dorsal Genital Nerve; Frequent bowel movements
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Electrical stimulation to the dorsal genital nerve.
  Interventions: Device: UCon

INTERVENTIONS:
Device: UCon — The participant self-administer electrical stimulation to the dorsal genital nerve (DGN) for 4 weeks using UCon

SUMMARY:
UCon is a medical device for treatment of the symptoms of overactive bladder and fecal incontinence (FI). It electrically stimulates the DGN through the skin to obtain modulated behaviour of the bladder/bowel musculature e.g., suppress undesired bladder/bowel activity to relieve the symptoms of the patient. This clinical investigation is designed as a single-arm, prospective, single-centre, early feasibility study.

DETAILED DESCRIPTION:
The overall purpose of the current clinical investigation is to evaluate the medical device (UCon) with respect to initial safety and device performance in a cohort of Spanish patients with FI over a treatment period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥ 18 years of age.
2. Participant is showing symptoms of FI.
3. Participant is able to communicate, provide feedback, understand and follow instructions during the course of the investigation, including using the device at home.

Exclusion Criteria:

1. Participant is medically unstable (acute illness or complication of a chronic condition that might affect the participants´ participation in the investigation).
2. Participant has an active infection in the genital area.
3. Participant has an implanted pacemaker, implantable drug pump or other active medical device (any medical device that uses electrical energy or other source of power to make it function).
4. Participant is pregnant, nursing or planning a pregnancy (to be confirmed with a negative pregnancy test). Women of childbearing potential must maintain effective contraception* during the interventional period judged by the investigator.
5. Participant is enrolled or planning to enrol in another clinical investigation or was enrolled in an investigational drug trial or medical device investigation within four weeks to enrolment.
6. Participant has neuropathy to a degree that is presumed to diminish the effect of the electrical stimulation, e.g., denervated patients and severe diabetic neuropathy.
7. Participant is currently receiving cancer treatment.
8. Participant has addictive behaviour defined as abuse of alcohol, cannabis, opioids, or other intoxicating drugs.
9. Participant does not speak and understand Spanish.

   * The following contraception is considered effective: Intrauterine device, hormonal contraceptives such as birth control pills, implants, contraceptive patch, vaginal ring, and contraceptive injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
PRIMARY SAFETY: To evaluate adverse events [initial safety] of UCon for treatment of the symptoms of FI in a home setting. | After 28 days (4 weeks)
  Characterization of adverse events and anticipated adverse device effects associated with the use of UCon during the investigational period.
PRIMARY PERFORMANCE: To evaluate the ratio of treatment change [performance] of FI symptoms in a home setting. | Change from baseline at 28 days (4 weeks) and 42 days (6 weeks)
  Ratio of subjects with at least 50% improvement of their FI symptoms from baseline. Participants shall complete an electronic bowel diary to report their symptoms

SECONDARY OUTCOMES:
SECONDARY SAFETY: To identify the number of subjects experiencing adverse events associated with the use of UCon during the investigational period. | After 28 days (4 weeks)
  Number of subjects experiencing adverse events and anticipated adverse device effects associated with the use of UCon.
SECONDARY PERFORMANCE: To evaluate whether subjects using UCon experience a change in their quality of life. | Change from baseline at 28 days (4 weeks) and 56 days (8 weeks, end of study)
  Ratio of subjects with a change in their self-reported quality of life measures as assessed by specific QoL questionnaires related to FI condition (St. Marks incontinence score and Rockwood Fecal Incontinence Quality of Life Scale). An overall score with greater values indicates a worse symptom outcome.
SECONDARY PERFORMANCE: To evaluate the ratio of subject that accept UCon and DGN stimulation [Device and treatment acceptability of UCon]. | After 28 days (4 weeks)
  Ratio of subjects that accept UCon and DGN stimulation as assessed by a satisfaction survey recorded after each stimulation period.

CONTACTS AND LOCATIONS:
Overall Officials: Eloy Espin Basany, MD, Principal Investigator — Vall d'Hebron University Hospital, 119, 08035 Barcelona, Spanien
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Spain